CLINICAL TRIAL: NCT04625218
Title: Hydroxychloroquine for the Treatment of SARS-CoV2 (COVID 19) in the Critically Ill Patient: Pharmacokinetic Study. (CHLORO-VID)
Brief Title: Hydroxychloroquine for the Treatment of SARS-CoV2 (COVID 19) : Pharmacokinetic Study
Acronym: CHLORO-VID
Status: Withdrawn | Type: Observational
Why Stopped: Hydroxychloroquine is not yet used for the Treatment of SARS-CoV2 (COVID 19)
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0155; 2020-A01094-35 (Other: IDRCB)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Pneumonia
Keywords: SARS-CoV-2; hydroxychloroquine; pharmacokinetics; bronchoalveolar lavage fluid; Intensive Care Unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples from D1 to Day 9 of the hydroxychloroquine treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, observational, open, monocentric multisite, pharmacokinetic study of hydroxychloroquine in critically ill patients. The aim of this study is to assess the pharmacokinetic behavior of hydroxychloroquine in COVID-19 critically ill patients treated with crushed hydroxychloroquine tablets (administered enterally using a nasogastric tube).

DETAILED DESCRIPTION:
Based on the in vitro activity against SARS-CoV-2 and preliminary clinical data, hydroxychloroquine is currently used in the management of COVID-19 patients. In the meantime, the efficacy as well as the dosage of hydroxychloroquine is highly debated. Because of the severity of COVID-19 and the pharmacokinetics of hydroxychloroquine in systemic lupus erythematosus patients, a loading dose was rapidly included in the new hospital regimens to optimize drug distribution in tissues and more precisely in the lungs. Due to the lack of information on the plasma/blood concentrations required to induce a virological/clinical effect, plasma/blood concentration is monitored in many European countries for patients whether or not they are included in clinical research protocols. This problem of relationship between efficacy and exposure is important in the critically ill patient because both the bioavailability and the variability of the pharmacokinetic parameters are potentially responsible for variations in concentrations.

This study is a prospective, observational, open, multisite, pharmacokinetics study of hydroxychloroquine in critically ill patients. There is no supplemental intervention or additional samples compared to the standard care of these patients in our teaching hospital. The total duration of the study is that of the duration of hospitalization in intensive care. The duration of the pharmacokinetic study is 9 days, starting on D1 of the treatment with hydroxychloroquine, and ending with the last recommended residual plasma control. The total duration of treatment with hydroxychloroquine is 10 days, as recommended by the High Council of Public Health in its opinion of March 23, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Hospitalized in intensive care, intubated and ventilated
* With COVID-19 pneumonia confirmed by Rt-PCR,
* Having as specific treatment hydroxychloroquine, whatever the dosage regimen
* Having had the monitoring of the residual concentrations carried out by the Pharmacokinetics and Toxicology Laboratory of the Federative Institute of Biology of the Toulouse University Hospital the clinical Pharmacology and Toxicology laboratory of the Toulouse University Hospital
* Person affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Minor patients
* Patients refusing to participate in the study
* Person participating in another research including an exclusion period still in progress.
* Contraindications to hydroxychloroquine: pre-existing retinopathy, known hypersensitivity to 4-aminoquinolines, hemolytic anemia, porphyria, G6PD deficiency, myasthenia gravis, association with citalopram, escitalopram, hydroxyzine, domperidone and piperaquine
* Patients undergoing treatment with medicines known to prolong the QT interval or likely to induce a cardiac arrhythmia such as for example anti-arrhythmics of class IA and III, tricyclic antidepressants and certain anti-infectives (in particular antibiotics of the family of macrolides and fluoroquinolones as well as trimethoprim-sulfamethoxazole).
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
residual plasma concentration | Day 3
  residual plasma concentration measured before re-administration of the treatment
residual plasma concentration | Day 5
  residual plasma concentration measured before re-administration of the treatment
residual plasma concentration | Day 7
  residual plasma concentration measured before re-administration of the treatment
residual plasma concentration | Day 9
  residual plasma concentration measured before re-administration of the treatment

SECONDARY OUTCOMES:
The number of days without artificial ventilation | Day 28
  number of days without artificial ventilation
The length of hospital stay in intensive care | Day 28
  The length of hospital stay in intensive care measured in days number
Survival | Day 28
  Statu alive or death
Viral replication in the control bronchoalveolar lavage fluid on Day 7 | Day 7
  Viral replication on Day 7 measured by biological analysis of the bronchoalveolar lavage fluid
Viral replication in the control bronchoalveolar lavage fluid on Day 14 | Day 14
  Viral replication on Day 14 measured by biological analysis of the bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie RUIZ, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France